CLINICAL TRIAL: NCT02198716
Title: Multi-centre, Randomised,Prospective Trial of Xience or Vision Stent, Management of Angina in the Elderly
Brief Title: Xience or Vision Stent Management of Angina in the Elderly
Acronym: XIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Adam de Belder, Consultant Cardiologist, Brighton and Sussex University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 2.0 20.06.2008
Record Dates: First submitted 2014-07-16; First posted 2014-07-24 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Elderly; Angina
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug eluting stent (Other): Percutaneous coronary intervention
  Interventions: Procedure: Percutaneous Coronary Intervention using drug eluting stents
- Bare Metal Stent (Other): Percutaneous Coronary Intervention
  Interventions: Procedure: Percutaneous Coronary Intervention using bare metal stents

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention using drug eluting stents — Percutaneous Coronary Intervention using drug eluting stents
  Other Names: Xience Drug eluting stent
  Arms: Drug eluting stent
Procedure: Percutaneous Coronary Intervention using bare metal stents — Percutaneous Coronary Intervention using bare metal stents
  Other Names: Vision BM stent
  Arms: Bare Metal Stent

SUMMARY:
The treatment of complex coronary disease causing limiting symptoms of angina with drug-eluting stent technology will prove superior to bare metal stent technology, with respect to a combined endpoint of mortality, MI, requirement for target vessel revascularisation and severe haemorrhage, in patients aged 80 or above.

ELIGIBILITY:
Inclusion Criteria:

* AGE>80
* Stable angina or acute coronary syndrome
* Coronary narrowing suitable for stenting that is either ≥15mm long and/or ≤3mm diameter.
* Any lesion with high risk of restenosis eg chronic total occlusion, bifurcation, severe calcification
* Any left main stem lesion

Exclusion Criteria:

* Acute ST segment elevation myocardial infarction
* Cardiogenic shock
* Platelet count =50 x 109/mm3
* Patient life expectancy < 1 year
* Known allergies to clopidogrel, aspirin, heparin, stainless steel, IV contrast or stent drug elutant
* Recent major GI haemorrhage (within 3 months)
* Any previous cerebral bleeding episode
* Participation in another investigational drug or device study
* Patient unable to give consent
* Clinical decision precluding the use of drug eluting stent

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 800 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Death/ Myocardial Infarction/Target Vessel Failure/Major Haemorrhage | 1 year
  This is a composite outcome measure consisting of multiple measures of the events of Death, Myocardial Infarction,Target Vessel Failure, and/or Major Haemorrhage

SECONDARY OUTCOMES:
Angina status | 1 year
  This will be assessed in two ways:
  i) by interview according to the Canadian Cardiovascular Society classification
  ii) by patient self-assessment using the Seattle questionnaire
Antianginal medication | 1 year
  This will be assessed using a single point scoring system, where a point is scored for each of the following:
  Nitrate (sublingual or spray) used 1 or mnore times during week prior to question Nitrate (oral) beta-blocker Calcium antagonist Use of Nicorandil
Procedural success | 1 Year
  Defined as TIMI 3 flow and <30% stenosis in the main vessel and TIMI 3 flow in the side branch
MACE (major adverse cardiovascular events) | 1 year
  Defined as death, myocardial infarction, or emergency (within 24 hours) coronary artery bypass grafting.
In-hospital complications | 1 Year
  Major procedural complications include Death Myocardial infarction Emergency coronary artery bypass surgery Stroke Bleeding ('Thrombolysis In Myocardial Infarction)
  Minor procedural complications include Ventricular rhythm disorder (tachy or brady) requiring intervention (e.g defibrillation, DC cardioversion or temporary pacing) Bleeding Pseudoaneurysm requiring compression or surgery Vascular access complication extending hospital stay by 1 or more night Transient ischaemic attack Wire loss or fracture Stent loss Undeployed stent detachment from balloon
Procedural cost | 1 Year
  The difference in procedural cost will be assessed using a composite of the number of, guidewires, balloons and stents opened or used and procedural time. Prolonged hospital stay is a further potential cost pressure in this age group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac Research Unit, Brighton, Sussex, United Kingdom